CLINICAL TRIAL: NCT04319471
Title: Single Arm, Open, Multicenter Phase II Clinical Study of Sufficient Chemotherapy Combine With Maintenance Chemotherapy in the Treatment of Oligometastatic Nasopharyngeal Carcinoma
Brief Title: Sufficient Chemotherapy Combine With Maintenance Chemotherapy in the Treatment of Oligometastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Jiangxi Provincial Cancer Hospital (Other); Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC003.1
Record Dates: First submitted 2020-03-22; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Maintenance Chemotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sufficient Chemotherapy Combine With Maintenance Chemotherapy (Experimental): Patients with oligometastatic Nasopharyngeal Carcinoma was given S-1 40-60mg bid d1-14, q4w, oral maintenance chemotherapy for 1 year or capecitabine 2500mg/m2/d twice daily oral d1-14, q4w after receiving sufficient chemotherapy and consolidative local therapy
  Interventions: Drug: Capecitabine/S-1; Drug: Chemotherapy; Radiation: Head and neck radiotherapy; Other: Local Consolidative Therapy

INTERVENTIONS:
Drug: Capecitabine/S-1 — Drug: Capecitabine/S-1
  Other Names: Maintenance chemotherapy
Drug: Chemotherapy — Gemcitabine (1000mg/m2) D1 D8+ nidaplatinum (80-100mg/m2) D2 q3w ×4-6cycle
Radiation: Head and neck radiotherapy — IMRT is uesd for the synchronous oligometastatic Nasopharyngeal Carcinoma；
Other: Local Consolidative Therapy — radiotherapy，surgery or interventional therapy for all metastatic sites.

SUMMARY:
This study is a randomized, phase II, prospective, multicenter clinical trial to evaluate the efficacy and safety of sufficient chemoradiotherapy plus oral capecitabine/S-1 for 1 year in the treatment of oligometastatic Nasopharyngeal Carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients with oligometastatic nasopharyngeal carcinoma (newly diagnosed or after treatment) ; patients with first diagnosis of nasopharyngeal carcinoma diagnosed by pathological biopsy; metastatic focus in principle need biopsy pathological diagnosis; but if the patient refuses to take the metastatic biopsy, the clinician decides with clinical evidence
2. Patients with a ECOG score of 0,1 or 2 and an expected survival period of more than 6 months; those who can cooperate in observing adverse reactions and outcomes;
3. At least one tumor lesion can be measured according to recist 1.1 criteria
4. Have good organ function
5. Informed consent signed and dated indicating that the patient has been informed of all relevant aspects of the study ;
6. Patients who are willing and able to comply with visiting arrangements, treatment plans, laboratory tests, and other research procedures ;
7. Be willing to comply with arrangements during the study to no longer participate in any other clinical studies related to drugs and medical devices.

Exclusion Criteria:

1. Patients with severe history of rapid-onset allergy to any of the drugs used in this study ;
2. Patients with local and/or regional recurrence;
3. Combine with other malignancies in 5 years (except non-melanin skin cancer or pre-invasion cervical cancer);
4. Any of the following conditions existed during the first six months of screening: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery transplantation, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism. patients known to have coronary artery disease, congestive heart failure that does not meet the above criteria or left ventricular ejection fraction < 50% and must use an optimized stable medical protocol determined by the therapist, if appropriate, to consult a cardiologist ;
5. Active infections, including tuberculosis, hepatitis b, hepatitis c, and human immunodeficiency virus. Patients with hbv surface antigen (hbsag) positive but HBV DNA <1000 copies/ml are eligible to participate in the study ;
6. Idiopathic pulmonary fibrosis, drug-induced pneumonia, organic pneumonia (bronchiolitis obliterans),Chest CT scans showing evidence of active pneumonia during history or screening of idiopathic pneumonia;
7. Substance abuse or alcohol addiction
8. Inability or limitation of civil capacity ;
9. Patients with physical or mental disorders who, according to the researchers, can not fully or fully understand the possible complications of the study ;
10. May increase the risk associated with the treatment of the study protocol, or may interfere with the interpretation of the study results and (as judged by the researchers) may render the patient unfit to participate in other severe acute or chronic medical conditions (including immune colitis, inflammatory bowel disease, non-infectious pneumonia, pulmonary fibrosis) or mental disorders (including dementia and epilepsy, recent, past year or active suicidal ideation or behavior) or laboratory abnormalities ;
11. Patients with expected survival <6 months ;
12. Previous diagnosis of immunodeficiency or known Human Immunodeficiency Virus (HIV) or acquired immunodeficiency syndrome (aids)-related diseases ;
13. Male or female pregnant or lactating women who have fertility but are unwilling or unable to use contraception throughout the study period and at least one year after the treatment programme ;
14. Large amounts of glucocorticoids or other immunosuppression have been used within 4 weeks of treatmen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival(PFS) | 12 months and 24 months
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.

SECONDARY OUTCOMES:
overall survival(OS) | 12 months and 24 months
  OS was defined as the time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Department of radiation oncology, Fujian cancer hospital, Fuzhou, Fujian, China